CLINICAL TRIAL: NCT04724876
Title: Meningitis Encephalitis: a Metagenomics-Based Etiology & Epidemiology Research (MEMBER Research)
Brief Title: Meningitis Encephalitis: a Metagenomics-Based Etiology & Epidemiology Research
Acronym: MEMBER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other); Air Force Military Medical University, China (Other); Peking Union Medical College Hospital (Other); The Second Hospital of Hebei Medical University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Chinese PLA General Hospital (Other); Xuanwu Hospital, Beijing (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Shandong Provincial Hospital (Other Government); Fudan University (Other); West China Hospital (Other); Henan Provincial People's Hospital (Other); Central South University (Other); The First Affiliated Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Jia Wei Wang,MD,PhD, MD, PhD, Professor, Beijing Tongren Hospital
Other Study IDs: TRECKY2020-141
Record Dates: First submitted 2020-12-08; First posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Central Nervous System Infections and Inflammations
MeSH Terms: conditions — Central Nervous System Infections; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — whole blood; serum; cerebrospinal fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Autoimmune encephalitis (AE) is caused by abnormal immune response mediated by autoimmune antibodies of patients, which can be detected by a serial of autoimmune antibodies[4,5,6,7]. At present, the traditional infection diagnosis mainly relies on microbial culture method, which has the characteristics of long cycle, high cost, low detection rate and complex detection process. About 30-60% of encephalitis have unknown etiology[2,3]. On the other hand, the diagnosis and classification of noninfectious encephalitis mainly depend on the detection of autoimmune antibodies, the scope of diagnosis and differential diagnosis is limited, and the relationship between autoimmune encephalitis and infection factors is still unclear. Metagenomics sequencing (mNGS) is a new method that does not rely on microbial culture and can directly detect pathogenic nucleic acids. It has the characteristics of fast, accurate, high throughput, no preference for different pathogen detection, and can detect known and unknown pathogens at the same time. Nowadays, mNGS is widely used in the field of pathogen detection.

ELIGIBILITY:
Inclusion Criteria:

* Either meet the items of 1, 2 or 1, 3

  1. The patient's age >14 years old, acute or subacute onset (less than 3 months), (first onset, treatment with anti-infection drugs and/or immunotherapy ≤5 days);
  2. The patient has the following symptoms:

     1. Dysmnesia,
     2. Seizures,
     3. Mental disorders,
     4. Abnormal behavior,
     5. Unconsciousness or coma,
     6. Dyskinesia or involuntary movement,
     7. lalopathy or be reticent,
     8. Dysphagia, sleep disorders, or autonomic nervous dysfunction,
     9. Ataxia.
  3. Patients with meningeal irritation sign, intracranial hypertension and other manifestations, satisfy at least 3 of the following symptoms:

     1. Headache,
     2. Fever,
     3. Stiff neck,
     4. Disturbance of consciousness,
     5. Kernig sign or brudzinski sign was positive.

Exclusion Criteria:

* 1. Patients with suspected metabolic encephalopathy and toxic encephalopathy have the above manifestations,
* 2. Patients with central nervous system tumor (primary or metastatic) have the above manifestations,
* 3. The patient with non-organic mental illness,
* 4. Patients who had undergone brain surgery within 6 months have the above symptoms after operation,
* 5. Patients with traumatic brain injury have the above manifestations,
* 6. Febrile convulsions caused by non-cerebral causes,
* 7. Patients with above manifestations due to other reasons such as cerebrovascular disease, genetic disease, etc;
* 8. Patients who refuse lumbar puncture or have contraindications to lumbar puncture;
* 9. Patients who withdraw informed consent.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected central nervous system infection.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-12-31 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
To elucidate the etiology and epidemiology of CNS infection all around China | within 2 weeks
  The Investigators use mNGS method to describe central nervous system infection spectrum.

CONTACTS AND LOCATIONS:
Overall Officials: Jiawei Wang, Doctor, Principal Investigator — Beijing Tong Ren Hospital
Locations (1):
- Beijing Tongren Hospital,Capital Medical University, Beijing, Beijing Municipality, China